CLINICAL TRIAL: NCT05137522
Title: Chidamide Combines With Etoposide and Methylprednisolone in the Treatment of Hemophagocytic Lymphohistiocytosis
Brief Title: Chidamide Combines With VP-16 and Methylprednisolone in the Treatment of HLH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chidamide,VP-16,HLH
Record Dates: First submitted 2021-11-24; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-08

CONDITIONS: Chidamide; Hemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Etoposide; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Chidamide combines with VP-16 and methylprednisolone
  Interventions: Drug: Chidamide combines with VP-16 and methylprednisolone

INTERVENTIONS:
Drug: Chidamide combines with VP-16 and methylprednisolone — Chidamide 30mg TIW po，etoposide 100 mg/m2 was administered day1; methylprednisolone 2mg/kg days 1 to 3,then 0.75mg/kg day 4 to 6，0.25mg/kg day 7 to 9，and 0.1mg/kg day 10 to 21

SUMMARY:
Chidamide combines with VP-16 and methylprednisolone in HLH

DETAILED DESCRIPTION:
This study aimed to investigate the efficacy and safety of Chidamide together with Etoposide and methylprednisolone for hemophagocytic lymphohistiocytosis

ELIGIBILITY:
Inclusion Criteria:Meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria; patients were diagnosed with EBV associated HLH (EBV-HLH) and lymphoma associated HLH.Age ≥18 years old, gender is not limited. Serum creatinine ≤ 1.5 times normal；NT-proBNP ≤ normal；Informed consent obtained.

-

Exclusion Criteria: Active bleeding of the internal organs or patients with new thrombotic diseases；Allergic to Chidamide and etoposide；Participate in other clinical research at the same time；HIV , HBV and HCV infected patients (HIV antibody positive)；History of QT interval prolongation, atrioventricular block, ventricular tachycardia, coronary atherosclerotic heart disease；Pregnant or lactating women and patients of childbearing age who refuse to take appropriate contraceptive measures during this trial. If the patient was male, he refused to use adequate contraceptive methods or donate semen during the study period and within 3 months after receiving the last cycle of drug study；patients judged by the investigator to be unsuitable to participate in this study.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment response | 4 weeks after Chidamide combines with VP-16 and methylprednisolone was used
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.Overall response rate (ORR) is defined as the ratio of patients with CR and PR to overall patients

SECONDARY OUTCOMES:
EBV-DNA copies | 4 weeks after Chidamide combines with VP-16 and methylprednisolone was used
  EBV-DNA copies in peripheral blood for patients with EBV positive when they enrolled
relapsed rate of HLH | 4 weeks after Chidamide combines with VP-16 and methylprednisolone was used
the response rate of lymphoma | 4 weeks after Chidamide combines with VP-16 and methylprednisolone was used
  lymphoma associated HLH

OTHER OUTCOMES:
treatment-related adverse events as assessed by CTCAE v5.0 | 4 weeks after Chidamide combines with VP-16 and methylprednisolone was used
  Adverse events including liver function damage, myelosuppression, infection, bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Wang Zhao, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China